CLINICAL TRIAL: NCT04519567
Title: A Phase 1 Multiple Ascending Dose Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Subcutaneous CTI-1601 Versus Placebo in Subjects With Friedreich's Ataxia
Brief Title: Multiple Ascending Dose Study of CTI-1601 Versus Placebo in Subjects With Friedreich's Ataxia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Larimar Therapeutics, Inc. (Industry)
Collaborators: Veristat, Inc. (Other); Metrum Research Group, LLC (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLIN-1601-102
Record Dates: First submitted 2020-08-17; First posted 2020-08-19 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Friedreich Ataxia
MeSH Terms: conditions — Friedreich Ataxia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CTI-1601 (Experimental)
  Interventions: Biological: CTI-1601
- Placebo (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: CTI-1601 — CTI-1601 is a recombinant fusion protein and is intended to deliver human frataxin, the protein deficient in Friedreich's ataxia
  Arms: CTI-1601
Biological: Placebo — Placebo Comparator
  Arms: Placebo

SUMMARY:
To evaluate the safety and tolerability of multiple ascending doses of CTI-1601 in participants with Friedreich's ataxia

DETAILED DESCRIPTION:
Multiple Ascending Dose (MAD), Double-Blind, Placebo Controlled Study.

To evaluate the safety and tolerability of multiple ascending doses of CTI-1601 in subjects with Friedreich's ataxia.

Secondary Objectives:

1. To evaluate the pharmacokinetics (PK) of CTI-1601 following, multiple, increasing, doses of subcutaneously (SC) administered CTI-1601.
2. To evaluate the pharmacodynamics (PD) of CTI-1601 following, multiple, increasing, doses of SC administered CTI-1601.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has genetically confirmed Friedreich's ataxia diagnosis manifested by homozygous GAA repeat expansions, with repeat sizing (if available) included on diagnostic report.
2. Subject is male or female, 18 years of age or older at screening
3. Subject must have a mFARS_neuro score ≥ 20 and be able to traverse a distance of 25 feet with or without some assistive device (cane, walker, crutches, self-propelled wheelchair) and (a) be able to sit upright with thighs together and arms crossed without requiring support on more than two sides; (b) be able to transfer from bed to chair independently or with assistance if, in the opinion of the principal investigator, the degree of physical disability does not result in undue risk to the subject while participating in the study; and (c) perform basic daily care, such as feeding themselves and personal hygiene, with minimal assistance.
4. Subjects must weigh > 40 kilograms (kg).

Exclusion Criteria:

1. Subjects who had a serious adverse event (SAE), an adverse event (AE) that is Grade 3 or higher according to the Common Terminology Criteria for Adverse Events (CTCAE), version 5.0 (or higher), or an AE considered clinically significant during participation in CLIN-1601-101 (NCT04176991).
2. Subjects who are confirmed as compound heterozygous (GAA repeat expansion on only one allele) for Friedreich's ataxia.
3. Subject use of investigational drug (other than CTI-1601) or device within 90 days prior to screening.
4. Subject requires use of amiodarone.
5. Subject used erythropoietin, etravirine, or gamma interferon within 3 months prior to screening.
6. Subject use of daily biotin supplementation that exceeds 30 mcg/day, either as part of a multivitamin or as a standalone supplement, within 7 days prior to study drug administration and/or throughout the entire study.
7. Subject has clinically significant arrhythmia on electrocardiogram (ECG), or evidence of predisposition to significant ventricular arrhythmia on ECG, or evidence of active and unstable coronary artery disease.
8. Male subject who has a QT interval corrected for heart rate using Fridericia's formula (QTcF) > 450 milliseconds or female subject who has a QTcF > 470 milliseconds on an ECG.
9. Subject has a screening echocardiogram left ventricular ejection fraction < 45 percent.
10. Subject has a history of aspiration, aspiration pneumonia, or recurrent episodes of pneumonia (greater than or equal to 2 episodes of pneumonia) within the last 12 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2020-07-31 (Actual); Primary Completion 2021-03-16 (Actual); Study Completion 2021-03-16 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Treatment Emergent Adverse Events | Through study completion, an average of 75 days
  Overall summary of Participants with Treatment Emergent Adverse Events
Number of Participants with Treatment Emergent Adverse Events by System Organ Classification and Preferred Term | Through study completion, an average of 75 days
  Overall summary of Participants with Treatment Emergent Adverse Events by System Organ Classification (MedDRA version 23.0)

SECONDARY OUTCOMES:
Pharmacokinetics - Maximum observed plasma concentration after multiple doses | At baseline and up to 15 days
  Summary assessment of changes in the maximum observed plasma concentration after multiple doses
Pharmacokinetics - Minimum or "trough" plasma concentration after multiple doses | At baseline and up to 15 days
  Summary assessment of minimum or "trough" observed plasma concentration after multiple doses just prior to the administration of a subsequent dose
Pharmacokinetics - Area under the concentration time curve (AUC) from time 0 through the last measurable time point | At baseline and up to 15 days
  Summary assessment of changes in the AUC from time 0 to the last measurable time point and during the dosing interval
Pharmacokinetics - Terminal half-life estimation | At baseline and up to 15 days
  Summary assessment of changes in the terminal half-life estimation
Changes from Baseline in Frataxin Levels in Buccal Cell | At baseline and up to 43 days
  Summary assessment of changes in frataxin levels in buccal cells
Changes from Baseline in Levels of Protein Markers in Buccal Cell | At baseline and up to 43 days
  Summary assessment of changes in levels of protein markers in buccal cells
Changes from Baseline in Gene Expression in Buccal Cells | At baseline and up to 43 days
  Summary assessment of changes in gene expression in buccal cells
Changes from Baseline in Frataxin Levels in Platelets | At baseline and up to 13 days
  Summary assessment of changes in frataxin levels in platelets
Changes from Baseline in Gene Expression in Whole Blood | At baseline and up to 16 days
  Summary assessment of changes in gene expression in whole blood
Changes from Baseline in Frataxin Levels in Skin Punch Cells | At baseline and up to 13 days
  Summary assessment of changes in frataxin levels in skin punch cells
Changes from Baseline in Levels of Defined Protein Markers in Blood | At baseline and up to 16 days
  Summary assessment of changes in levels of defined protein markers in blood
Changes from Baseline in Levels of Specialized Lipids in Blood | At baseline and up to 16 days
  Summary assessment of changes in levels of specialized lipids in blood

CONTACTS AND LOCATIONS:
Overall Officials: Magdy Shenouda, M.D., Principal Investigator — Clinilabs, Inc.
Locations (1):
- Clinilabs Drug Development Corporation, Eatontown, New Jersey, United States

REFERENCES:
- [Background] Koeppen AH. Friedreich's ataxia: pathology, pathogenesis, and molecular genetics. J Neurol Sci. 2011 Apr 15;303(1-2):1-12. doi: 10.1016/j.jns.2011.01.010. PMID 21315377
- [Background] Delatycki MB, Corben LA. Clinical features of Friedreich ataxia. J Child Neurol. 2012 Sep;27(9):1133-7. doi: 10.1177/0883073812448230. Epub 2012 Jun 29. PMID 22752493
- [Background] Goodkin DE, Hertsgaard D, Seminary J. Upper extremity function in multiple sclerosis: improving assessment sensitivity with box-and-block and nine-hole peg tests. Arch Phys Med Rehabil. 1988 Oct;69(10):850-4. PMID 3178453
- [Background] Rudick R, Antel J, Confavreux C, Cutter G, Ellison G, Fischer J, Lublin F, Miller A, Petkau J, Rao S, Reingold S, Syndulko K, Thompson A, Wallenberg J, Weinshenker B, Willoughby E. Clinical outcomes assessment in multiple sclerosis. Ann Neurol. 1996 Sep;40(3):469-79. doi: 10.1002/ana.410400321. PMID 8797541
- [Background] Plasterer HL, Deutsch EC, Belmonte M, Egan E, Lynch DR, Rusche JR. Development of frataxin gene expression measures for the evaluation of experimental treatments in Friedreich's ataxia. PLoS One. 2013 May 17;8(5):e63958. doi: 10.1371/journal.pone.0063958. Print 2013. PMID 23691127
- See also: Friedreich's Ataxia Research Alliance — http://www.curefa.org/